CLINICAL TRIAL: NCT01021800
Title: Modulation of the Immune Response in Patients With Pancreatic Tubular Adenocarcinoma
Acronym: SYSTHER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blood Transfusion Centre of Slovenia (Other Government)
Responsible Party: Primoz Rozman, MD PhD, Blood Transfusion Centre of Slovenia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-11

CONDITIONS: Pancreatic Tubular Adenocarcinoma
Keywords: Pancreatic tubular adenocarcinoma adjuvant setting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cell infusion (Experimental)
  Interventions: Biological: MIS

INTERVENTIONS:
Biological: MIS — Cell infusion

SUMMARY:
Interventional study of modulation of immune response in patients with pancreatic tubular adenocarcinoma after resection and gemcitabine treatment. When included, patients are pre-treated with moderate doses of cyclophosphamide. Then infusions of allogeneic mononuclear cells are given.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2 at the time of inclusion
* Following R0 or R1 pancreatic tubular adenocarcinoma resection and adjuvant gemcitabine treatment

Exclusion Criteria:

* Pregnancy
* Less than 3 mths expected survival
* Serious comorbidity
* Age above 70 yrs

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
PROGRESSION FREE SURVIVAL | 1 YEAR

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Department for Gastroenterolgy, Ljubljana, Ljubljana, Slovenia